CLINICAL TRIAL: NCT06741514
Title: A Clinical Benefits Survey Study of Precice Intramedullary Limb Lengthening System (IMLL) Limb Lengthening Procedures
Brief Title: A Study of Precice Intramedullary Limb Lengthening System (IMLL) Limb Lengthening Procedures
Status: Enrolling by invitation | Type: Observational
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Other Study IDs: NUVA.ILL0923
Record Dates: First submitted 2024-11-07; First posted 2024-12-19 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Limb Length Discrepancy
Keywords: Precice; limb lengthening; limb lengthening discrepancy; surgery; index bone; femur; tibia; limb length

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Parents or Legal Gaurdians: Parents or legal guardians of patients who were enrolled in the Precice IMLL arm of the retrospective data collection study (NUVA.IMLL0723).
  Interventions: Device: Precice IMLL

INTERVENTIONS:
Device: Precice IMLL — Parents or legal guardians of children that previously received the Precice IMLL will complete a survey. No additional or new interventions will be administered.

SUMMARY:
The Sponsor is conducting a survey to understand how parents or legal guardians feel about the benefits of using the Precice IMLL System to lengthen limbs in children who are 12 years old or younger.

DETAILED DESCRIPTION:
All participants in this survey study will be the parent or legal guardian of a child who previously underwent surgery for limb length discrepancy according to the practitioner's standard of care, was 12 years of age or younger at the time of surgery, and is enrolled in the Precice IMLL arm in protocol NUVA.IMLL0723. The parent or legal guardian will be familiar with the patient's preoperative and postoperative condition, surgical treatment, postoperative care, and clinical outcomes.

Each parent or legal guardian will complete the perceived clinical benefits survey questionnaire once. The survey will be administered as either a paper-based questionnaire via mail or over the phone or an electronic questionnaire completed via a secure online application.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for inclusion in this perceived clinical benefit survey study, the following inclusion criteria must be met:

  1. Participants must be a parent or legal guardian of a subject already enrolled in the Precice IMLL arm of the study, "A Retrospective Review of the Clinical and Radiographic Outcomes Following the Use of the Precice Intramedullary Limb Lengthening System (IMLL) in Pediatric Limb Lengthening Procedures" (NUVA.IMLL0723).
  2. The parent or legal guardian must be familiar with the patient's preoperative and postoperative condition, surgical treatment, postoperative care, and clinical outcomes.
  3. Informed consent from the parent or legal guardian of the patient is required for participation.

Exclusion Criteria:

* There are no exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Parents or legal guardians of patients who were enrolled in the Precice IMLL arm of the retrospective data collection study (NUVA.IMLL0723).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Perceived clinical benefits of the Precice Intramedullary Limb Lengthening (IMLL) Survey System | 1 year post-op
  Non-validated survey to assess the perceived clinical benefits of the Precice Intramedullary Limb Lengthening (IMLL) System in limb lengthening procedures in pediatric patients ages 12 years and younger as reported by parents or legal guardians.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs Study Director, Study Director — Globus Medical Inc
Locations (2):
- United States (2):
  - Paley Orthopedic and Spine Institute, West Palm Beach, Florida
  - Nationwide Childrens Hospital, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No